CLINICAL TRIAL: NCT03257293
Title: A Randomized Control Trial of a Modified Cystoscopy Method to Reduce Pain Perception
Brief Title: A Trial of a Modified Cystoscopy Method to Reduce Pain Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10016740
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Hematuria; Bladder Cancer; Bladder Disease
MeSH Terms: conditions — Hematuria; Urinary Bladder Neoplasms; Urinary Bladder Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Cystoscopy (Active Comparator)
  Interventions: Behavioral: Routine Cystoscopy
- Modified Cystoscopy (Experimental)
  Interventions: Behavioral: Modified Cystoscopy

INTERVENTIONS:
Behavioral: Modified Cystoscopy — The objective of this study is to examine whether a non-pharmacologic modification in procedure of cystoscopies improves patient perception of pain and discomfort.
  Arms: Modified Cystoscopy
Behavioral: Routine Cystoscopy — Routine cystoscopy as done as part of routine clinical practice
  Arms: Routine Cystoscopy

SUMMARY:
The goal of this project is to improve patient experience of cystoscopy using a non-pharmacologic modification of procedure. Cystoscopy is a common outpatient procedure for urology patients and is usually performed without sedation. However, there is limited research into reduction of patient discomfort throughout this procedure. The proposed modification technique was selected based on a well-documented psychological phenomenon in which only particular moments over the course of an aversive event determine the resultant perception of the experience. It is hypothesized that implementation of the technique will decrease the recalled pain intensity of the cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 undergoing cystoscopy for the first time for diagnostic investigation will be approached to participate in this study.

Exclusion Criteria:

* Cystoscopies involving other interventions concurrently (e.g. biopsy, urethral dilation, removal of ureteral stent, etc.) will be excluded.
* Patients currently taking medication for chronic pain (e.g. opioids, Tricyclic antidepressants (TCAs)) will be excluded from the study.
* Patients less than 18 years of age will be excluded.
* Patients who have received a cystoscopy previously will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Pain Experience rated on the visual analogue scale | 1 hour
  The primary outcome of the study will be pain experience, as rated on the visual analogue scale provided.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Power, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No